CLINICAL TRIAL: NCT01541735
Title: Effect of Pantoprazole on Insulin Secretion in Patients With Type 2 Diabetes
Brief Title: Pantoprazole on Insulin Secretion in Diabetes
Acronym: IBP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Manuel Gonzalez Ortiz, Principal Investigator, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IBP1301-93
Record Dates: First submitted 2012-02-20; First posted 2012-03-01 (Estimated); Results first posted 2014-02-21 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-01

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Insulin; Pantoprazole
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance | interventions — Pantoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo of calcined magnesia, capsules
  Interventions: Drug: placebo
- Pantoprazole (Experimental): The pantoprazole will be administered in 40mg capsules
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole — The pantoprazole will be administered in capsules of 40mg. The dose will be 1 capsule per day during 45 days.
  Other Names: Pantozol
  Arms: Pantoprazole
Drug: placebo — Placebo 40 mg dose.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the effect of pantoprazole on insulin secretion in drug-naïve patients with type 2 diabetes.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) has become a major health problem worldwide with a high prevalence and related mortality, and a high rate of disability in the economically active. In Mexico the prevalence was 14.4% reported one of the highest in Latin America and estimated a cost of $ 778 million allocated for this disease in 2010, i.e., the tenth place worldwide. Within its pathophysiology are alterations in the secretion and insulin action, qualitatively and quantitatively, which implies a challenge for long-term metabolic control with the pharmacological arsenal available today. Since the function of pancreatic β cell decreases as a function of time and lack of control is essential metabolic find drugs that can preserve pancreatic cell mass and even promote neogenesis, with the aim of restoring the physiological secretion of insulin have been lost in the early stages of type 2 diabetes to achieve optimal glycemic control sustained over time to avoid complications and reduce the costs associated with the disease.

Have been evaluated in animal models with promising results Proton Pumps Inhibitors (PPI) for the restoration of glucose and the preservation of pancreatic cell function, including promoting its growth through increased levels of gastrin, which appears to act as a growth factor. However, at present no such mechanisms have been evaluated in humans, it would be interesting to assess the effect of administration of a PPI such as pantoprazole is, on the phases of insulin secretion in patients with T2DM recent diagnosis.

Material and Methods: Randomized, double-blind, placebo controlled clinical trial. Population: 14 drug-naive adults patients with T2DM and obesity. Hyperglycemic-hyperinsulinemic clamp to assess the phases of insulin secretion. Intervention for 45 days: pantoprazole 40mg or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Drug-Naive
* No complications
* HbA1c 7 to < 9%
* Fasting plasma glucose < 210mg/dl
* Body mass index 30.0 to 39.9 and body weight stable for at least 3 months before the study
* Non smokers
* Blood pressure < 130/80

Exclusion Criteria:

* Diabetes complications
* Women pregnant or stage of lactation
* Hepatic, renal, autoimmune disease
* Take drugs with effects on insulin secretion
* Zollinger-Ellison disease
* Gastric or pancreatic tumor.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Gonzalez, PhD, Principal Investigator — Instituto Mexicano del Seguro Social. Centro Medico Nacional de Occidente. Unidad de Investigación Médica en Epidemiologia Clínica
Locations (1):
- Instituto Mexicano del Seguro Social. Hospital de Especialidades., Guadalajara, Jalisco, Mexico

REFERENCES:
- [Derived] Gonzalez-Ortiz M, Martinez-Abundis E, Mercado-Sesma AR, Alvarez-Carrillo R. Effect of pantoprazole on insulin secretion in drug-naive patients with type 2 diabetes. Diabetes Res Clin Pract. 2015 Apr;108(1):e11-3. doi: 10.1016/j.diabres.2015.01.039. Epub 2015 Feb 7. PMID 25704601

RESULTS

PARTICIPANT FLOW:
Groups:
- Pantoprazole: The pantoprazole will be administered in 40mg capsules PO, 30 minutes before to breakfast during 45 days
- Placebo: Placebo of calcined magnesia, capsules PO, 30 minutes before to breakfast during 45 days
Period: Overall Study
Arm/Group | Pantoprazole | Placebo
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pantoprazole | Placebo | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (7.1) | 46.2 (9.6) | 48.0 (8.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Mexico | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: First Phase of Insulin Secretion
Description: The hyperglycemic-hyperinsulinemic clamp technique is perform to assess the phases of insulin secretion: first, late and total insulin secretion.
Time Frame: Change from Baseline at 45 days. (plus or minus 3 days)
Population: The analysis was determined per protocol and sample size was calculated whit the formula for clinical trial
Measure: Mean (Standard Deviation); unit: µU/ml
Arm/Group | Pantoprazole | Placebo
Number analyzed (Participants) | 7 | 7
µU/ml | 13.8 (5.5) | 15.9 (9.3)

2. Secondary Outcome: Glycated Hemoglobin A1C
Time Frame: Change from Baseline in glycated hemoglobin A1C at 45 day.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Pantoprazole | Placebo
Number analyzed (Participants) | 7 | 7
percentage | 7.5 (.38) | 7.8 (.45)

3. Primary Outcome: Second Phase of Insulin Secretion
Description: Change from baseline in first phase insulin secretion at 45 day. (plus or minus 3 days)
Time Frame: Baseline and 45 day
Measure: Mean (Standard Deviation); unit: µU/ml
Arm/Group | Pantoprazole | Placebo
Number analyzed (Participants) | 7 | 7
µU/ml | 35.9 (21.2) | 38.4 (30.1)

4. Primary Outcome: Total Insulin Secretion
Description: The hyperglycemic-hyperinsulinemic clamp technique is performed to assess the total insulin secretion
Time Frame: Change from baseline of total insulin secretion at 45 day (plus or minus 3 days)
Measure: Mean (Standard Deviation); unit: µU/ml
Arm/Group | Pantoprazole | Placebo
Number analyzed (Participants) | 7 | 7
µU/ml | 29.0 (15.8) | 31.5 (23.4)

ADVERSE EVENTS:
Arm/Group | Pantoprazole | Placebo
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

LIMITATIONS AND CAVEATS:
The intervention time was short to evaluate a total change in the primary outcome variables

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No